CLINICAL TRIAL: NCT00067743
Title: A Multicenter, Open-Label Study to Evaluate the Preliminary Safety and Efficacy of CC-5013 in the Treatment of Complex Regional Pain Syndrome (CRPS)
Brief Title: A Study of CC-5013 in the Treatment of Complex Regional Pain Syndrome (CRPS)
Acronym: CRPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Donald Manning, MD, PhD, Vice President Clinical Research and Development, Celgene Corportation
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-CRPS-001
Record Dates: First submitted 2003-08-26; First posted 2003-08-27 (Estimated); Last update posted 2008-01-03 (Estimated); Status verified 2006-12

CONDITIONS: Complex Regional Pain Syndrome (RSD)
Keywords: Pain; Pain syndrome; Reflex sympathetic dystrophy; CC-5013; CC5013; Revlimid; Celgene; CRPS
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain; Somatoform Disorders; Reflex Sympathetic Dystrophy | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Open Label trial
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — supplied as 5 mg capsules. Dosing as directed by physician but to start at 10 mg per day
  Other Names: Revlimid

SUMMARY:
This is a multicenter, open-label study in adult subjects with Type 1 Complex Regional Pain Syndrome. Subjects diagnosed with unilateral Type 1 CRPS will be enrolled sequentially to receive CC-5013 10 mg/day orally. For each subject the study consists of two phases: Pre-treatment phase(1 wk) and treatment phase (12 wks)

DETAILED DESCRIPTION:
Once the subject completes the 12 week treatment phase the subject is eligible to continue on the trial. Subjects may continue until no further benefit is obtained.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Type 1 CRPS as defined by modified International Association for the Study of Pain criteria (App 1) for at least one year duration
* Unilateral involvement of a distal hand or foot with or without proximal speed must be present. The most severely affected limb will be designated the index limb.
* CRPS pain severity score in the index limb of 4 or greater on an 11-point (0-10) NRS (Appendix I).
* Opioid analgesics, non-opioid analgesics, non-steroidal anti-inflammatory drugs, anticonvulsants and antidepressant drugs may be continued provided that the subject was on stable doses for at least four weeks prior to the Treatment phase.
* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug.
* In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug.
* WCBP must agree to have pregnancy tests every 4 weeks while on study drug.
* The average CRPS pain severity score in the index limb at the end of the Pre-Treatment Phase I (must be 4 or greater) and 2 each of the daily scores over the week must be within +/- one point of this average.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Prior treatment with CC-5013
* Prior development of an allergic reaction/hypersensitivity while taking thalidomide.
* Prior development of a moderate or sever rash or any desquamation while taking thalidomide.
* Pregnant or lactating females.
* Active litigation, compensation or disability issues related to CRPS.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of the treatment phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-08; Primary Completion 2004-10 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety | throughout the trial

SECONDARY OUTCOMES:
Change in CRPS pain rating in index limb compared to baseline | throughtout trial compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Donald Manning, MD, PhD, Study Director — Celgene Corporation
Locations (6):
- United States (6):
  - UCSD Center for Pain and Palliative Medicine, La Jolla, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - UNC Hospitals University of North Carolina, Chapel Hill, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Swedish Pain Management, Seattle, Washington